CLINICAL TRIAL: NCT04018781
Title: Eval CONPARMED Haute-Bretagne : Guaranteeing the Continuity of the Care Pathway for the Elderly Patient: Evaluation of a Territorial Approach of Clinical Pharmacy
Brief Title: Guaranteeing the Continuity of the Care Pathway for the Elderly Patient: Evaluation of a Territorial Approach of Clinical Pharmacy
Acronym: CONPARMED
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30022; 2019-A00455-52 (Other: Id-RCB)
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Medication Reconciliation at Discharge
Keywords: Medication reconciliation; clinical pharmacy
MeSH Terms: interventions — Medication Reconciliation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MR group: Patients who benefit from a full process of medication reconciliation (entrance and discharge) before being discharged to home.
  Interventions: Other: medication reconciliation
- Control group: Patients who benefitted from a medication reconciliation at entrance only before being discharged to home.
  Interventions: Other: medication reconciliation

INTERVENTIONS:
Other: medication reconciliation — During hospitalization, the hospital pharmacist will carry out a pharmaceutical analysis for all patients included in the study, each time the prescription is changed and within a maximum of 24 hours (working days).
  If necessary, in consultation with the doctor in charge of the patient, the pharmacist may also propose a pharmaceutical interview to the patient at any time during his hospitalisation (e.g. proposal for the de-prescription of benzodiazepines, Proton Pump Inhibitors, etc., according to the recommendations in force).

SUMMARY:
In the context of the ageing of the French population, drug iatrogeny in the elderly is a major public health issue, responsible for approximately 7,500 deaths per year and 3.4% of hospitalizations among patients aged 65 and over.

The interest of the Medication Reconciliation (MR) in reducing medication errors and unintentional discrepancies in prescriptions at transition points in patients' medication care pathways no longer seems to be in doubt both in France and abroad.

On the other hand, the literature on the clinical impact of these drug errors (i. e. occurrence of an adverse drug event (ADE) or readmission rates) is currently limited in France and presents variable results abroad.

DETAILED DESCRIPTION:
The medication reconciliation implementation mobilizes human resources (pharmacists, pharmacy technician, nurses...) and constitutes an investment for healthcare institutions. However, the resulting improvement in patients' health status (and the potential reduction in ADEs) could reduce their care consumption and thus reduce costs from a healthcare system perspective. We therefore propose to assess the cost-effectiveness of this care strategy.

Finally, we will study the impact of the MR deployment on existing professional organizations, both in hospital and between community healthcare professionals and hospital as well as its conditions of implementation.

ELIGIBILITY:
Inclusion criteria :

* Patient > 65 years old
* Patient hospitalized inside one of the thirteen wards in the 6 hospitals participating in the study
* Informed consent given

Non inclusion and Exclusion Criteria :

* Patients in palliative care
* Persons deprived of their liberty

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years admitted inside one of the thirteen wards from 6 hospitals located around Rennes and Fougères, between 13/06/2019 and 13/09/2019
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Adverse drug event-related hospital revisits | 30 days after discharge
  Rate of adverse drug event-related hospital revisits within 30 days after discharge

SECONDARY OUTCOMES:
General Practitioner consultation | 30 days after discharge
  Rate of General Practitioner consultation within 30 days after discharge
All-causes readmissions and/or Emergency Department visits | 30 days after discharge
  Composite rate of readmissions and/or Emergency Department visits within 30 days after discharge
All-causes readmissions and/or Emergency Department visits | 90 days after discharge
  Composite rate of readmissions and/or Emergency Department visits within 90 days after discharge
Incremental Cost-Effectiveness Ratio (ICER) at Day 30 | 30 days after discharge
  Medico-economic analysis : Incremental Cost-Effectiveness Ratio (ICER) : cost per hospitalization for Drug Adverse Event avoided and cost per all-causes hospitalization, according to a collective perspective at Day 0.
Incremental Cost-Effectiveness Ratio (ICER) at Day 90 | 90 days after discharge
  Medico-economic analysis : Incremental Cost-Effectiveness Ratio (ICER) : cost per hospitalization for Drug Adverse Event avoided and cost per all-causes hospitalization, according to a collective perspective at Day 90.
Patient reported experience measures | 7 days after discharge
  Patient reported experience measures are realized by a short phone call interview, 7 days after the patients' homecoming
Severity of Unintended Medication Discrepancies | At admission
  Severity of Unintended Medication Discrepancies intercepted during medication reconciliation at admission
Number of Unintended Medication Discrepancies | At admission
  Number of Unintended Medication Discrepancies intercepted during medication reconciliation at admission
Impact of the implementation of the intervention on professional organizations | Before and after the implementation of the intervention in the participating wards
  Qualitative analysis based on :
  * First, an inventory of organizations prior to the implementation of the intervention in participating health facilities
  * Then, an assessment of the impacts of the implementation of the intervention on different aspects of professional organizations: collaborative exchanges, multi-professional information sharing, division of labour, exchanges with city practitioners, learning effects, evolution of professional practices.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit HUE, MD, PhD, Study Director — University Hospital of Rennes
Locations (6):
- France (6):
  - Hopital des Marches de Bretagne, Antrain
  - General Hospital, Fougères
  - General Hospital, Janzé
  - General Hospital, Montfort-sur-Meu
  - University Hospital, Rennes
  - General Hospital, Saint-Méen-le-Grand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bajeux E, Alix L, Cornee L, Barbazan C, Mercerolle M, Howlett J, Cruveilhier V, Line-Iehl C, Cador B, Jego P, Gicquel V, Schweyer FX, Marie V, Hamonic S, Josselin JM, Somme D, Hue B. Pharmacist-led medication reconciliation at patient discharge: a tool to reduce healthcare utilization? an observational study in patients 65 years or older. BMC Geriatr. 2022 Jul 13;22(1):576. doi: 10.1186/s12877-022-03192-3. PMID 35831783